CLINICAL TRIAL: NCT06827899
Title: A Multicenter, Prospective, Single-arm Clinical Study of Veneclax, Chidaniline Combined With Azacitidine (VCA) Followed by Decitabine + MAG Regimen (D-MAG) in the Treatment of Elderly Untreated Acute Myeloid Leukemia (AML)
Brief Title: Veneclax, Chidaniline Combined With Azacitidine Followed by Decitabine + MAG Regimen in the Treatment of Elderly Untreated AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: Fujian Provincial Hospital (Other); Fujian Cancer Hospital (Other Government); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Jieyang People's Hospital (Other); Huizhou Municipal Central Hospital (Other)
Responsible Party: Principal Investigator, Bing, Xu, The First Affiliated Hospital of Xiamen University, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-04
Record Dates: First submitted 2025-02-11; First posted 2025-02-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- veneclax, chidaniline combined with azacitidine (VCA) followed by decitabine + MAG regimen (D-MAG) (Experimental)
  Interventions: Drug: veneclax, chidaniline combined with azacitidine (VCA) followed by decitabine + MAG regimen (D-MAG)

INTERVENTIONS:
Drug: veneclax, chidaniline combined with azacitidine (VCA) followed by decitabine + MAG regimen (D-MAG) — Specified dose on specified days

SUMMARY:
A multicenter, prospective, single-arm clinical study of veneclax, chidaniline combined with azacitidine (VCA) followed by decitabine + MAG regimen (D-MAG) in the treatment of elderly untreated acute myeloid leukemia (AML)

DETAILED DESCRIPTION:
A multicenter, prospective, single-arm clinical study of veneclax, chidaniline combined with azacitidine (VCA) followed by decitabine + MAG regimen (D-MAG) in the treatment of elderly untreated acute myeloid leukemia (AML)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed acute myeloid leukemia (non-M3). Have not received treatment before and cannot accept standard cytarabine and anthracycline induction regimen treatment due to age or comorbidity or patient preference;
2. Age >= 60 years old, male or female, expected survival time greater than 3 months;
3. Estimated creatinine clearance >= 30 mL/min;
4. AST and ALT <= 3.0 x ULN (unless considered due to leukemic organ involvement). Bilirubin <= 1.5 x ULN (unless considered due to leukemic organ involvement);
5. ECOG <= 2;
6. Able to understand and voluntarily provide informed consent.

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL) and low-risk cytogenetics, such as t(8;21), inv(16), or t(16;16);
2. Active central nervous system leukemia;
3. A history of myeloproliferative neoplasms (MPN), including myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myelogenous leukemia (CML) with or without BCR-ABL1 translocation and AML with BCR- ABL1 translocation;
4. HIV-positive patients and/or HBV or HCV active infection (documented by HBV-DNA and HCV-RNA positive tests);
5. Suffering from chronic respiratory diseases requiring continuous oxygen inhalation, or having an obvious history of kidney, nervous system, psychiatric, endocrine, metabolic, immune, liver, and cardiovascular diseases;
6. Suffering from malabsorption syndrome or other diseases that exclude the enteral route of administration;
7. Clinically significant QTc interval prolongation (male > 450 ms; female > 470 ms), ventricular tachycardia and atrial fibrillation, second-degree heart block, myocardial infarction, and congestive heart failure within one year before enrollment patients, and patients with coronary heart disease who have clinical symptoms and need drug treatment;
8. Active, uncontrolled severe infection;
9. There is a history of other malignant tumors within 2 years, except for the following cases: adequately treated carcinoma in situ of the cervix or carcinoma in situ of the breast; basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
10. White blood cell count > 25 x 10^9/L (hydroxyurea or leukapheresis can meet this standard);
11. Mental disorders that will hinder research participation;
12. Participants have received the following treatments: hypomethylation agents, venetoclax and/or chemotherapy for myelodysplastic syndrome (MDS), solid organ transplantation;
13. Any other circumstances that the investigator believes that the patient is not suitable to participate in this trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 60 months
  Defined as the time interval from treatment initiation to the occurrence of induction failure, relapse, or death, whichever came first.

SECONDARY OUTCOMES:
Complete Remission (CR) rate | Up to 60 months
  The percent of participants with complete remission (CR) was defined in accordance with the IWG Response Criteria in AML.
Overall Survival (OS) | Up to 60 months
  OS will be measured from the date of registration to the date of the event (i.e., death) or the date of last follow-up to evaluate that event. Patients who are event-free at their last follow-up evaluation will be censored at that time point.
Overall Response Rate (ORR) | Up to 60 months
  Defined as the percentage of participants achieving a best overall response of complete response (CR), CR with incomplete blood count recovery (CRi), or partial response (PR).
General Health Status/Quality of Life | Up to 60 months
  Will be assessed by Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- Bing Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No